CLINICAL TRIAL: NCT06425393
Title: Prevalence and Risk Factors of Intrafamilial Helicobacter Pylori Infection in Hong Kong: a Prospective Cohort Study
Brief Title: Intrafamilial Helicobacter Pylori Infection in Hong Kong
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lily Wan Ying LAI, Resident doctor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024.143
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: H.Pylori Infection
Keywords: H.pylori infection

STUDY DESIGN:
Intervention Model Description: Patients who are diagnosed to have H. pylori infection by either histology, rapid urease test or urea breath test will be recruited. At least 1 household member of each H. pylori infected subject will also be recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H. pylori positive subjects (No Intervention): The H. pylori infected subject is responsible for providing details of the number of household members, family structure, family history of gastric diseases, family economy, living conditions, family hygiene and living habits. Patients also need to provide personal information including HKID, ethnicity.
- H. pylori positive subjects' household members (Experimental): The household members of the index subjects will be invited to complete a questionnaire which includes the baseline demographics, past medical history, personal hygiene and living habits. Also, they will be received urea beath test (UBT). Referral will be given to those positive result household members.
  Interventions: Diagnostic Test: Urea beath test (UBT)

INTERVENTIONS:
Diagnostic Test: Urea beath test (UBT) — H. pylori infection will be tested using a 13C-urea breath test Kit for all enrolled family members, following the manufacturer's instructions. The sensitivity and specificity of the assay are both over 95%, according to the manufacturer's introduction.
  Arms: H. pylori positive subjects' household members

SUMMARY:
It is a single-centre, prospective cohort study, which will be conducted in a tertiary academic hospital. The study aims to investigate intrafamilial H. pylori infection status and to identify risk factors for H. pylori infection among household members.

The rate of intrafamilial H. pylori spread in Hong Kong is currently unknown. It is also not clear whether the same risk factors for intrafamilial spread of H. pylori infection also apply in Hong Kong. In contrast to mainland China and Taiwan , recent consensus guideline on H. pylori management in Hong Kong in 2023 recommends against routine testing of asymptomatic household members or family members of H. pylori-infected adults. There is a knowledge gap on whether the family-based H. pylori screening is cost effective in our locality. Thus, the investigator aim to investigate infection status of household members of H. pylori infected individuals and risk factors for household infection in Hong Kong. The result from this study will shed light on the role of family-based screening and can inform future healthcare policy making on the strategy of H. pylori management and treatment in Hong Kong, ameliorating H. pylori infection-related disease and gastric cancer burden for society.

DETAILED DESCRIPTION:
Helicobacter pylori infects around half of the population in the world, and it is believed to affect more than half of population in Hong Kong. H. pylori infection is a well-known cause of chronic gastritis, peptic ulcer diseases and gastric cancer. Early detection and eradication of H. pylori infection is of utmost importance.

H. pylori infection is mainly transmitted by oral-oral, faecal-oral routes and water sources . Emerging studies demonstrated that intrafamilial spread is common. Recent national, family-based epidemiological study on H. pylori infection in mainland China showed a high familial infection rate ranging from 50.27% to 85.06%. In another study in central China, it was found that all family members were infected with H. pylori in 27.8% of the H. pylori infected households. Therefore, detection and eradication of H. pylori infection in family are very important to prevent development of H. pylori related diseases. Instead of the traditional strategies for individual-based management of H. pylori infection like 'test and treat' and 'screen and treat' strategies, a new strategy 'family- based H. pylori infection control and management' has been introduced. In 2021, China published a consensus report on the Family-based H. pylori infection control and management with an aim to reduce intrafamilial H. pylori spread in the Chinese population. In Taiwan, where the incidence of GC is high, a preventive strategy with 13C-urea breath test screening using the index case method and outreach the family members of the positive index cases. Eradication therapies for those who test positive and to follow up 2 years later to test the reinfection rate has been implemented to reduce the incidence of gastric cancers and reduce the cancer health inequality in indigenous communities.

Previous studies have identified several risk factors for intrafamilial transmission of H. pylori infection. Large family size of 3 or more in a household and living in highly infected areas in Northwest China were risk factors for household H. pylori infection while family members with higher income and education level , using serving spoons or chopsticks , drinking boiled water from tap source were associated with lower risk of household infection.

There is concern on the re-infection rate of H. pylori after eradication therapy. A systemic review revealed that global annual recurrence, reinfection and recrudescence rates of H. pylori were 4.3% (95%CI: 4-5), 3.1% (95%CI: 2-5) and 2.2% (95%CI: 1-3), respectively. An observational study in Turkey found that for H. pylori infected patients with whole family testing and eradication, the recurrence rate was 7.1% 9 months after treatment. On the other hand, when only the infected patient was eradicated but the whole family infection was not treated, the recurrence rate was 38.6% 9 months after treatment. These results suggest that treatment of the whole infected family is of great value in controlling H. pylori re-infection and preventing recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adults age>=18 years of age
* For H. pylori infected patients only: Diagnosed to have H. pylori infection by either histology, rapid urease test or urea breath test
* Written informed consent obtained

Exclusion Criteria:

* Unable to perform urea breath test
* Contraindications for urea breath test
* Used antibiotics within the past month/proton pump inhibitors within two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-11 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Rate of H. pylori infection in household members | during the study period, 2 years
  The rate of H. pylori infection in household members of H. pylori infected subjects from the given UBT

IPD SHARING:
Plan to Share IPD: No
There will be no plan to share individual participant data.